CLINICAL TRIAL: NCT02188225
Title: Comparison of the Effects of Acupuncture and Fluoxetine on Quality of Life in Menopausal Women
Brief Title: Comparison of Acupuncture and Fluoxetine on Quality of Life in Menopausal Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Gonabad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Narjes Bahri, Instructor of midwifery education, Gonabad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GMU.REC.1393.56
Record Dates: First submitted 2014-07-10; First posted 2014-07-11 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Hot Flash; Quality of Life
Keywords: Hot flash; Acupuncture; Fluoxetine; Quality of life
MeSH Terms: conditions — Hot Flashes | interventions — Acupuncture Therapy; Fluoxetine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture (Experimental): 12 sessions of acupuncture / 3 sessions weekly/ 20 minutes each session
  Interventions: Procedure: acupuncture
- fluoxetine (Active Comparator): 10 mg daily
  Interventions: Drug: fluoxetine

INTERVENTIONS:
Procedure: acupuncture — 12 sessions acupuncture during 12 weeks (3 sessions weekly), each session lasting 20 minutes
  Other Names: Manual acupuncture
  Arms: Acupuncture
Drug: fluoxetine — 10 mg/ daily
  Other Names: flouxetine
  Arms: fluoxetine

SUMMARY:
The purpose of this study is to comparison the effect of acupuncture and Fluoxetine on improvement quality of life among menopausal women.

DETAILED DESCRIPTION:
This clinical trial is designed in two arm include acupuncture and fluoxetine group to evaluate the effect of these intervention on improvement quality of life among menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Last menstrual cycle 12 months ago
* natural menopause
* 4 episodes of hot flash daily
* follicle stimulating hormone (FSH)= 30-110 IU/L , E2<18pg/ml
* thyroid-stimulating hormone(TSH)= 0.4-4/0 IU/ml
* No using of herbal agent for treatment of hot flash
* having score in Beck depression Inventory<10
* No existence of any medical problems and using drugs

Exclusion Criteria:

* Not completing all acupuncture sessions
* Not completing fluoxetine admission
* Withdraw the study

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2014-07; Primary Completion 2019-02-20 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life in menopausal women | 3 months after start sampling
  Quality of life using MENQOL questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Narjes Bahri, PhD Student, Principal Investigator — Gonabad University of Medical Sciences
Locations (2):
- Iran (2):
  - Gonabad University of Medical Sciences, Gonābād, Khorasan Razavi
  - Narjes Bahri, Mashhad, Razavi Hkorasan Privience

IPD SHARING:
Plan to Share IPD: Undecided